CLINICAL TRIAL: NCT02051322
Title: Comparison of Lung Administration With Three Different Nebulizer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trunk
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Jet Nebulizer (Experimental): Nebulization with a jet nebulizer and a classic mask
  Interventions: Device: Jet Nebulizer
- Trunk Mask Nebulizer (Experimental): Nebulization with a je nebulizer and a trunk mask
  Interventions: Device: Trunk Mask Nebulizer
- Aerobika Nebulizer (Experimental): Nebulization with an Aerobika
  Interventions: Device: Aerobika Nebulizer

INTERVENTIONS:
Device: Jet Nebulizer
  Arms: Jet Nebulizer
Device: Trunk Mask Nebulizer
  Arms: Trunk Mask Nebulizer
Device: Aerobika Nebulizer
  Arms: Aerobika Nebulizer

SUMMARY:
Comparison between three modalities of nebulization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects

Exclusion Criteria:

* Pulmonary disease
* Cardiac disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Lung deposition by urinary measure | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium